CLINICAL TRIAL: NCT00756691
Title: A Radiopharmacokinetic and Radiodosimetric Phase I Imaging Study of 18F-FAZA
Status: Withdrawn | Type: Observational
Why Stopped: Limited scanner availability
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: PK-FAZ-003
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hypoxic Tumours
Keywords: 18F-FAZA; Positron Emission Tomography; Radiation dosimetry; Pharmacokinetics
MeSH Terms: interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: First 5 consecutive 18F-FAZA avid subjects that undergo up to 5 PET scans, 13 blood and 2 urine samples over 4.5 hours
  Interventions: Other: 18F-FAZA
- 2: Next 5 consecutive 18F-FAZA avid subjects that undergo up to 4 PET scans, 8 blood and 2 urine samples over 5.5 hours
  Interventions: Other: 18F-FAZA

INTERVENTIONS:
Other: 18F-FAZA — Radioactive dose of 110-600 MBq per injection. A single pre-treatment injection of 18F-FAZA will be permitted per patient

SUMMARY:
Hypoxia (little of no oxygen) is considered to be an important characteristic of a patient's tumour that may help predict patient outcomes and/or help inform patient management decisions. 18F-FAZA Positron Emission Tomography (PET) can detect hypoxic tumours because 18F-FAZA accumulates in hypoxic tissues. This study is being done to learn more about the processes by which 18F-FAZA is absorbed, distributed, metabolized (built-up and broken down) and eliminated by the body.

DETAILED DESCRIPTION:
A Phase I Radiopharmacokinetic and Radiodosimetric study of 18F-FAZA. Prior to treatment, subjects will receive a single injection of 18F-FAZA. Subjects will undergo a series of 5-5 PET scans, and will have 8-13 blood samples and 2 urine samples taken at specified time points over a 4.5-5.5 hour period. 18F-FAZA PET images will be reviewed to develop a dynamic uptake model, and blood and urine samples will be analyzed for unchanged 18F-FAZA and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Male of Female > or = to 18 years of age. If female of child-bearing potential and outside of the window of 10 days since the first day of the last menstrual period, a negative pregnancy test required
* Subjects with known primary or suspected metastatic SCC head and neck; NSCLC; SCLC; GBM; lymphoma, or NET with at least one lesion > 1 cm in diameter
* Able and willing to follow instructions and comply with the protocol
* Provide written informed consent prior to participation in the study
* Karnofsky Performance Scale Score of 70-100

Exclusion Criteria:

* Previous treatment for their primary or metastatic SCC head and neck, NSCLC, SCLC, GBM, Lymphoma, or NET
* Bilirubin > or = to 200 umol/L
* Creatinine > or - to 150 umol/L
* AST or ALT > or = to 5 times the upper limits of normal
* Serious medical conditions such as: congestive heart failure, unstable angina, unstable ventricular arrhythmia, uncontrolled psychiatric conditions, serious infections, uncontrolled diabetes
* Nursing or pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known primary or suspected metastatic carcinoma of the following: squamous cell carcinoma (SCC) of the head and neck, small (SCLC) and non-small cell lung cancer(NSCLC), Glioblastoma multiforme (GBM), lymphoma, or neuroendocrine tumours (NET).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To Collect imaging-based data for radiopharmacokinetic and radiodosimetric analyses. | 2 years

SECONDARY OUTCOMES:
To determine radiation dosimetry and optimal imaging times | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MB, FRCPC, Principal Investigator — Professor, Department of Oncology